CLINICAL TRIAL: NCT03944005
Title: A Randomized Controlled Double Blinded Multicentre Study Comparing Discharge Readiness of Combined Adductor Canal and IPACK Blocks to LIA for Knee Arthroplasty Surgery.
Brief Title: Comparing Two Regional Anesthesia Interventions for Knee Arthroplasty.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to achieve funding and logistic issue due to COVID.
Sponsor: Western University, Canada (Other)
Collaborators: George Eliot Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Abhijit Biswas, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113078
Record Dates: First submitted 2019-01-29; First posted 2019-05-09 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Knee Arthroplasty
Keywords: knee arthroplasty; discharge readiness; analgesia; adductor canal block; ipack; LIA
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): Spinal Anesthesia + ACB continuous catheter+ iPACK + Sham LIA
  Interventions: Procedure: Spinal Anesthesia + ACB continious catheter + iPACK + Sham LIA
- Comparator Group (Sham Comparator): Spinal Anesthesia + LIA + Sham Blocks
  Interventions: Procedure: Spinal Anesthesia + LIA + Sham Blocks

INTERVENTIONS:
Procedure: Spinal Anesthesia + ACB continious catheter + iPACK + Sham LIA — ACB - On identification of adductor canal,10ml ropivacaine 0.5% with 1:400,000 epinephrine will be injected to surround the femoral artery.Following catheter placement, another 10ml of the same solution will be injected. Continuous infusion of 5ml/hr 0.2% ropivacaine will be infused till considered ready to discharge.
  Ipack - Posterior knee infiltration will be performed following ACB. On visualization of femoral condyle and popliteal artery, 20ml ropivacaine 0.5% with 1:400,000 epinephrine will be infiltrated in muscular space between popliteal artery and posterior femoral condyle.
  Spinal anesthesia will be performed following nerve blocks. All patients will receive 2-3ml of 0.75% preservative-free bupivacaine at the level of L2-3 or L3-4 intervertebral space.
  LIA - Patients in Group 1 will receive local infiltration 100ml of normal saline around the knee capsule of 100ml of normal saline by the surgeons as a Sham injection.
  Arms: Study Group
Procedure: Spinal Anesthesia + LIA + Sham Blocks — ACB - On identification of adductor canal, 10ml of saline as a sham solution will be injected to surround the femoral artery. Following catheter placement, another 10ml of the same solution will be injected. Continuous infusion of 5ml/hr of saline will be infused till considered ready to discharge.
  Ipack - Posterior knee infiltration will be performed following ACB. On visualization of the femoral condyle and popliteal artery, 20ml of saline will be infiltrated in the muscular space between popliteal artery and posterior femoral condyle.
  Spinal anesthesia will be performed following the nerve blocks. All patients will receive 2-3ml of 0.75% preservative-free bupivacaine injected at the level of L2-3 or L3-4 intervertebral space.
  LIA - Patients will receive local infiltration by the attending surgeon intraoperatively with 300mg of ropivacaine (100ml of 0.3% ropivacaine),30 mg of ketorolac, and 10mg of morphine around the knee capsule.
  Arms: Comparator Group

SUMMARY:
Osteoarthritis of the knee is a common disease of the elderly and knee arthroplasty is indicated in severe cases to improve long term pain and function. Along with perioperative quality analgesia, functional recovery is paramount in the postoperative period.Loco-regional techniques provide effective analgesia and can mitigate several side effects of systemic opioids administration. Also, adequate motor sparing analgesia( to prevent weakness of the thigh muscle) following total knee arthroplasty (TKA) is therefore paramount to ensure effective rehabilitation, early recovery, readiness to discharge or timely hospital discharge.

There are several motor sparing regional technique described in literature. Adductor canal block (ACB), use of intrathecal ( IT) morphine and local infiltration by the surgeons (LIA) are such examples. Previous studies have shown the combination of ACB and IT morphine to be superior than LIA in providing analgesia.

Posterior knee infiltration (IPACK), involves blocking the branches of the tibial nerve which provides sensory innervation for the posterior aspect of the knee. In combination with ACB, a motor sparing analgesic intervention is possible for knee arthroplasty.

Rationale for doing the study is to evaluate

1. The effectiveness of IPACK block as a part of multimodal analgesic approach to knee arthroplasty surgery.
2. Enhanced recovery from superior motor sparing analgesia.
3. early hospital discharge We hypothesize that, following total knee arthroplasty surgery, the combination of continuous adductor canal catheter and I-PACK blocks will achieve a decrease in the time to readiness to hospital discharge as measured by the following four criteria: (1) adequate analgesia; (2) independence from intravenous opioids; (3) ability to independently stand, walk 3 m (metres), return, and sit down; and (4) independently ambulate 30 m without limitation of time. We postulate this will occur by providing superior motor-sparing analgesia compared to LIA for knee arthroplasty surgery.

DETAILED DESCRIPTION:
Introduction Osteoarthritis of the knee is a common disease of the elderly and knee arthroplasty (TKA) is indicated in severe cases to improve long term pain and function. Inadequate perioperative pain control is a strong predictor of persistent pain beyond 3 months.

Analgesic modalities for TKA Several analgesia regimes exist for TKA. Multimodal regimens including both loco-regional techniques or systemic analgesics. Loco-regional techniques provide effective analgesia and can mitigate the side effects of systemic opioids including nausea and vomiting, pruritus, respiratory depression and urinary retention.

Muscle weakness following regional anesthesia technique may induce fall, hinder early rehabilitation and prolong hospitalization. Motor sparing analgesic (do not cause weakness of muscles) are in vogue due to enhance early rehabilitation and analgesia. Local Infiltration Analgesia (LIA), Adductor Canal Block (ACB) and posterior infiltration of the knee (IPACK) are examples of motor sparing interventions utilized for TKA surgery.

LIA involves the injection of high volumes of dilute local anesthetic solution directly into the articular and peri-articular tissues during the surgical procedure.

ACB consists on the administration of local anesthetic in the adductor canal, an aponeurotic compartment in the mid-thigh containing the femoral vessels and several distal branches of the lumbar plexus that contribute to the innervation of the anterior aspect of the knee.

Posterior knee infiltration (IPACK), involves ultrasound guided injection of local anesthetics in the muscular plane between the popliteal artery and the femoral condyles. This involves blocking the branches of the tibial nerve which provides sensory innervation for the posterior aspect of the knee Hypothesis We hypothesize that, following total knee arthroplasty surgery, the combination of continuous adductor canal catheter and IPACK blocks will achieve a decrease in the time to readiness to hospital discharge as measured by the following four criteria: (1) adequate analgesia; (2) independence from intravenous opioids; (3) ability to independently stand, walk 3 m(metres),return and sit down; and (4) independently ambulate 30 m without limitation of time. We postulate this will occur by providing superior motor-sparing analgesia compared to LIA for knee arthroplasty surgery.

Methodology. This will be a multicentric Randomized controlled double blinded study. Proposed timeline is three years following ethics approval.

Study Centre The study will take place in two university hospitals; University Hospital, London Health Sciences Centre, London, Ontario and George Elliot Hospital, Warwickshire, United Kingdom. These centers have the clinical volume, technical expertise equipment setup, previous experience in this area of research, and research support needed to carry out the proposed study.

Research Ethics Board (REB) Approval An application has been submitted to the University Health Network, Western University and Leister University Ethics Board for REB approval Informed Consent Patients will be identified from operation schedule list from the surgical secretaries office a month in advance of their operation.An information package containing a letter of introduction, study information and consent form will be posted to the patients address as mentioned in power chart a month in advance of OR schedule. Then the patient we will contacted by our study team over phone to introduce the study and verbal consent. Written consent will happen on the day of admission. The investigator will be a physician and will not be participating in the patient's care on the day of surgery.

Patients will be informed of the procedures involved in the study, the chances of being assigned to one of the 2 groups, the risks and benefits of participating, and of their right to withdraw from the study at any time without adversely affecting their clinical care. The investigators will retain a signed, witnessed consent form. The telephone number of the chair of the George Elliot Hospital Research Board and Western University Research Ethics Board will be provided to study participants to contact for information on the rights of human subjects participating in clinical research.

Blinding A Pharmacist not directly involved in patient care will prepare all study drugs. The patient, anesthesiologist performing the block and looking after the patient in the block operating room, surgeons, physiotherapists and the investigator collecting outcome data will be unaware of study group allocation. The documentation in the anesthetic chart will be written as study interventions instead of the actual procedure.

Randomization and study groups

Study participants will be randomly allocated to one of two groups using a computer-generated list of random numbers and sealed opaque envelopes using Lawson Redcap. The study groups will receive the following interventions:

Group 1. Spinal Anesthesia + ACB continuous catheter+ IPACK + Sham LIA (100 ml of normal saline infiltrated by the surgeons at the end of surgery) Group 2. Spinal Anesthesia + LIA + Sham Blocks(20 ml of normal saline ACB and continuous infusion+ IPACK each) Interventions and Peri-operative management ACB and continuous catheter placement. ACB will be performed prior to surgery in the block room. Monitoring of vital signs will include non-invasive blood pressure, electrocardiogram, and pulse oximetry. Supplemental oxygen will be administered. After performing a "time-out" procedure including verification of "correct surgical site", sedation will be achieved with IV Midazolam in 1 mg increments and IV Fentanyl in 25 mcg increments as needed. Ultrasound examination of the thigh will be performed using a high frequency linear probe (5-12 MHz range) with either a Philips Sparq or Sonosite Turbo. The study participants will be positioned supine with the operative knee slightly flexed and the hip externally rotated. Under sterile technique, the adductor canal will be identified as an aponeurotic compartment limited by the sartorius muscle antero-medially, the adductor muscles posteriorly and the vastus medialis muscle laterally. After skin infiltration of 1 - 3 ml of 2% lidocaine, a 80 mm, 22 gauge, short-bevel echogenic needle (Sonoplex, Pajunk, Norcross, Georgia, Arrow depending on the institution) will be advanced, in plane with the ultrasound beam in the mid-thigh, at equal distance from the groin and the patella. 10ml of study solution will be injected to surround the femoral artery and the catheter would be placed in the adductor canal lateral to the artery. After the placement of the catheter, another 10 ml of the study solution will be injected. Continuous infusion of 5mls/hr of 0.2% of ropivacaine will be infused till considered ready to discharge. For Group 1 the active study drug will consist of 20ml of ropivacaine 0.5% with 1:400,000 epinephrine. In Group 2, study participants will receive 20ml of 0.9% saline as a bolus and 5mls/hr of normal saline infusion in the postoperative period.

IPACK Posterior knee infiltration will be performed following ACB. The study participants will remain supine with knee flexed and internally rotated. After full asepsis, the ultrasound probe will be placed on the superior- lateral surface of the knee joint. On visualization of the femoral condyle and popliteal artery, an infiltration of the drug will be made in the muscular space between the popliteal artery and the posterior femoral condyle. Group 1 receive 20ml of ropivacaine 0.5% with 1:400,000 epinephrine while Group 2 will receive 20ml of 0.9%saline.

Spinal Anesthesia with IT morphine Spinal anesthesia will be performed following the ACB and IPACK per standard institutional practice. The study participants will be placed in the sitting position and a 25-gauge Whitacre needle will be introduced at the L2-3 or L3-4 intervertebral levels to enter the intrathecal space under aseptic condition. All patients will receive 2-3 ml of 0.75% preservative-free bupivacaine.

Local Infiltrative Analgesia (LIA) For they study participants in group 2, the knee joint will be infiltrated by the surgeon intraoperatively with 300 mg of ropivacaine (100 ml of 0.3% ropivacaine),30 mg of ketorolac, and 10mg of morphine. Study Participants in Group 1 will receive local infiltration of 100ml of normal saline as a Sham injection.

Post-operative Systemic Analgesics

Standardized perioperative systemic analgesics will be provided to all subjects following current standard institutional practice. This will include:

1. Acetaminophen 3 to 4 g orally daily for 5 days,
2. Celecoxib 100 to 200 mg orally twice a day (or an alternate non-steroidal anti-inflammatory drug for those with sulfa allergy),
3. Hydromorphone 1-2 mg/morphine 5-10 mg/oxycodone 5-10 mg (or equivalent) orally every two hours as needed.

Intravenous patient-controlled analgesia with hydromorphone or morphine at equivalent doses will be prescribed as a "rescue" modality to be started only if oral analgesics fail to achieve a pain score of less than 5 as is standard institutional practice. Patients will be followed twice daily by the Acute Pain Service team who will be unaware of study group allocation and will make changes to the analgesic regimen as required by the clinical situation.

Sample Size Calculation Based of local data, the investigators hypothesize that the intervention, for a total of 532 participants (266 per group) the investigators will be able to detect a 20% difference in (length of stay)LOS from 2.8 days to 2.24 days. Based on this effect size, an alpha of 0.05 and a beta of 0.2, an estimate of sample size to be 532 (266 patients per group) was calculated.

Statistical Analysis Normality of continuous outcomes will be assessed visually (using histograms of raw and/or transformed data) and numerically (using the Shapiro-Wilk test). If the raw or transformed data are approximately normally-distributed, then a parametric method (t test) will be used for analysis, otherwise a non-parametric or semi-parametric method will be used (0.5 quantile [median] regression for non-time-to-event data and Cox regression for time-to-event data). Data will be presented as mean, standard deviation (SD) or median/ interquartile range (IQR). 95% confidence interval (CI) for the differences between groups will be constructed using standard techniques (for normally distributed outcomes) or using bootstrapping of 10,000 replications (for non-normally distributed outcomes).

Categorical outcomes will be analyzed using Fisher's exact test, along with the relative risk and its two-sided 95% CI. We will perform regression adjustment for any prognostically important differences between groups in baseline variables. A P value of < 0.05 will be considered significant.

Data Monitoring Committee Two researchers from the department of Anesthesia, Dr. Craig Railton and Dr. Mahesh Naggapa will form Data Monitoring Committee. They will meet once a year to review the results and advice the PI accordingly. None of the members of the Data Monitoring Committee will be involved in any other way with the conduct of the trial, except the routine, blinded intra or postoperative care of the study participants.

Confidentiality and DATA sharing All information gathered during the course of the study will be stored in a secure, locked filing cabinet, in a locked office of principal investigator. A master list with patient identification information (name, birth date, surgeon and surgical date) will be maintained separately from a deidentified list. This will allow for review of pertinent information if required. When entering and analyzing data, only study subject identification numbers will be used to ensure patient confidentiality. All personal identification data will be kept in the study regulatory binder, separate from study data. Study results will be presented in a way that makes it impossible to identify individual participants. The data will be collected in institutional REDCAP accounts and shared within institution. Data analysis will be performed by the LHSC Group.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status I-III
* 18 -70 years of age
* BMI 18 - 40
* Scheduled for elective unilateral primary total knee arthroplasty under spinal anesthesia.
* Able to ambulate independently with a standard wheeled walker as maximum mobility aid.

Exclusion Criteria:

* Revision knee arthroplasty
* Bilateral knee arthroplasty
* Inability to provide informed consent
* Patient scheduled for a second knee arthroplasty operation at a later date.
* Neuropathic pain or sensory disorders of the surgical limb already diagnosis by a physician.
* Contraindication to regional anesthesia.
* Chronic opioid use defined as > 60 mg of daily oral morphine equivalents.
* Patients who did not receive spinal anesthesia with intrathecal morphine or needed general anesthetics due to failed spinal anesthesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Time to achieve a collective four-point criterion for readiness to discharge from hospital after knee arthroplasty surgery. | 3 days
  1- adequate analgesia - pain score less than 4 on numerical rating scale of 11. (0 signifies no pain and 10 signifies maximum possible pain). Assessment will be performed in postoperative care unit (PACU) and every 12 hours till hospital discharge.
  2 - independence from intravenous opioids. Assessment will be performed in postoperative care unit (PACU) and every 12 hours till hospital discharge.
  3 - ability to independently stand, walk 3 metres (m), return and sit down (TUG test). Assessment will be performed every 12 hours till hospital discharge.
  4 - independently ambulate 30m with or without mechanical support (crutch) without any time limit. Assessment will be performed every 12 hours till hospital discharge.

SECONDARY OUTCOMES:
Post-Operative pain scores | 3 days
  Pain will be assessed on a 11 point numerical scale of '0' to '10'. Zero signifies no pain whereas 10 signifies maximum pain. Pain score will be evaluated during the preoperative assessment, on admission to PACU after surgery and every 12 hours in the postoperative period until discharge. Analysis will be performed as cumulative 24-hour pain score till discharge as area under the curve analysis. Pain scores will be measure at rest and movement
Total opioid consumptions in I.V. morphine equivalents | 3 days
  Total opioid consumptions in I.V. morphine equivalents on admission to PACU (postoperative care unit) after surgery and daily until discharge
Functional outcomes | 3 days and at 3rd month
  The functional outcome measures will consist of the TUG test and WOMAC score. The TUG test will be done in post-operative period only when the physiotherapists certify the patient is capable of mobilization. The test will be performed once during the pre-operative assessment period and then every 12 hour in the postoperative period until readiness to discharge is achieved. Other functional outcomes measured will be range of knee motion in the postoperative period and distance moved at a time on every postoperative day at physiotherapy assessment. WOMAC score will be evaluated over the phone after three months of recovery, will be assessed over phone. They will be called after 3 months, with permission from the patient, next of kin or family doctor.
Total length of hospital stay | 3 days
  Actual hospital length of stay in days after surgery, irrespective of readiness to discharge.
Nausea and vomiting | 3 days
  Nausea and Vomiting needing medication for treatment
Pruritus | 3 days
  Pruritus -needing medication for treatment
Respiratory Distress | 3 days
  3. Respiratory distress - needing emergency/immediate assessment by the attending physician
urinary retention | 3 days
  Retention of urine needing catheterization.

CONTACTS AND LOCATIONS:
Locations (2):
- London Health Sciences Centre, London, Ontario, Canada
- George Elliot Hospital NHS Trust, Nuneaton, Warwickshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Plan to publish/share the aggregate summary of the results instead of individual patient data. Individual patient's de-identified results could be shared depending on journal requirement at the time on publication.

REFERENCES:
- [Background] Zhang XL, Cheng T, Zeng BF; Chinese Medical Association; Chinese Orthopaedic Association. Experts' consensus on minimally invasive surgery for total joint arthroplasty. Orthop Surg. 2011 Aug;3(3):147-51. doi: 10.1111/j.1757-7861.2011.00134.x. No abstract available. PMID 22009643
- [Background] Puolakka PA, Rorarius MG, Roviola M, Puolakka TJ, Nordhausen K, Lindgren L. Persistent pain following knee arthroplasty. Eur J Anaesthesiol. 2010 May;27(5):455-60. doi: 10.1097/EJA.0b013e328335b31c. PMID 20299989
- [Background] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Background] Johnson RL, Kopp SL, Hebl JR, Erwin PJ, Mantilla CB. Falls and major orthopaedic surgery with peripheral nerve blockade: a systematic review and meta-analysis. Br J Anaesth. 2013 Apr;110(4):518-28. doi: 10.1093/bja/aet013. Epub 2013 Feb 24. PMID 23440367
- [Background] Wasserstein D, Farlinger C, Brull R, Mahomed N, Gandhi R. Advanced age, obesity and continuous femoral nerve blockade are independent risk factors for inpatient falls after primary total knee arthroplasty. J Arthroplasty. 2013 Aug;28(7):1121-4. doi: 10.1016/j.arth.2012.08.018. Epub 2012 Dec 21. PMID 23265274
- [Background] Ilfeld BM, Mariano ER, Girard PJ, Loland VJ, Meyer SR, Donovan JF, Pugh GA, Le LT, Sessler DI, Shuster JJ, Theriaque DW, Ball ST. A multicenter, randomized, triple-masked, placebo-controlled trial of the effect of ambulatory continuous femoral nerve blocks on discharge-readiness following total knee arthroplasty in patients on general orthopaedic wards. Pain. 2010 Sep;150(3):477-484. doi: 10.1016/j.pain.2010.05.028. Epub 2010 Jun 22. PMID 20573448
- [Background] Machi AT, Sztain JF, Kormylo NJ, Madison SJ, Abramson WB, Monahan AM, Khatibi B, Ball ST, Gonzales FB, Sessler DI, Mascha EJ, You J, Nakanote KA, Ilfeld BM. Discharge Readiness after Tricompartment Knee Arthroplasty: Adductor Canal versus Femoral Continuous Nerve Blocks-A Dual-center, Randomized Trial. Anesthesiology. 2015 Aug;123(2):444-56. doi: 10.1097/ALN.0000000000000741. PMID 26079800
- [Background] Sztain JF, Machi AT, Kormylo NJ, Abramson WB, Madison SJ, Monahan AM, Khatibi B, Ball ST, Gonzales FB, Sessler DI, Mascha EJ, You J, Nakanote KA, Ilfeld BM. Continuous Adductor Canal Versus Continuous Femoral Nerve Blocks: Relative Effects on Discharge Readiness Following Unicompartment Knee Arthroplasty. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):559-67. doi: 10.1097/AAP.0000000000000279. PMID 26115189
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Terkawi AS, Mavridis D, Sessler DI, Nunemaker MS, Doais KS, Terkawi RS, Terkawi YS, Petropoulou M, Nemergut EC. Pain Management Modalities after Total Knee Arthroplasty: A Network Meta-analysis of 170 Randomized Controlled Trials. Anesthesiology. 2017 May;126(5):923-937. doi: 10.1097/ALN.0000000000001607. PMID 28288050
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Essving P, Axelsson K, Kjellberg J, Wallgren O, Gupta A, Lundin A. Reduced hospital stay, morphine consumption, and pain intensity with local infiltration analgesia after unicompartmental knee arthroplasty. Acta Orthop. 2009 Apr;80(2):213-9. doi: 10.3109/17453670902930008. PMID 19404806
- [Background] Vendittoli PA, Makinen P, Drolet P, Lavigne M, Fallaha M, Guertin MC, Varin F. A multimodal analgesia protocol for total knee arthroplasty. A randomized, controlled study. J Bone Joint Surg Am. 2006 Feb;88(2):282-9. doi: 10.2106/JBJS.E.00173. PMID 16452738
- [Background] Sawhney M, Mehdian H, Kashin B, Ip G, Bent M, Choy J, McPherson M, Bowry R. Pain After Unilateral Total Knee Arthroplasty: A Prospective Randomized Controlled Trial Examining the Analgesic Effectiveness of a Combined Adductor Canal Peripheral Nerve Block with Periarticular Infiltration Versus Adductor Canal Nerve Block Alone Versus Periarticular Infiltration Alone. Anesth Analg. 2016 Jun;122(6):2040-6. doi: 10.1213/ANE.0000000000001210. PMID 27028771
- [Background] Sogbein OA, Sondekoppam RV, Bryant D, Johnston DF, Vasarhelyi EM, MacDonald S, Lanting B, Ganapathy S, Howard JL. Ultrasound-Guided Motor-Sparing Knee Blocks for Postoperative Analgesia Following Total Knee Arthroplasty: A Randomized Blinded Study. J Bone Joint Surg Am. 2017 Aug 2;99(15):1274-1281. doi: 10.2106/JBJS.16.01266. PMID 28763413
- [Background] Biswas A, Perlas A, Ghosh M, Chin K, Niazi A, Pandher B, Chan V. Relative Contributions of Adductor Canal Block and Intrathecal Morphine to Analgesia and Functional Recovery After Total Knee Arthroplasty: A Randomized Controlled Trial. Reg Anesth Pain Med. 2018 Feb;43(2):154-160. doi: 10.1097/AAP.0000000000000724. PMID 29315129
- [Background] Burckett-St Laurant D, Peng P, Giron Arango L, Niazi AU, Chan VW, Agur A, Perlas A. The Nerves of the Adductor Canal and the Innervation of the Knee: An Anatomic Study. Reg Anesth Pain Med. 2016 May-Jun;41(3):321-7. doi: 10.1097/AAP.0000000000000389. PMID 27015545
- [Background] Anagnostopoulou S, Kostopanagiotou G, Paraskeuopoulos T, Chantzi C, Lolis E, Saranteas T. Anatomic variations of the obturator nerve in the inguinal region: implications in conventional and ultrasound regional anesthesia techniques. Reg Anesth Pain Med. 2009 Jan-Feb;34(1):33-9. doi: 10.1097/AAP.0b013e3181933b51. PMID 19258986
- [Background] Davis JJ, Bond TS, Swenson JD. Adductor canal block: more than just the saphenous nerve? Reg Anesth Pain Med. 2009 Nov-Dec;34(6):618-9. doi: 10.1097/AAP.0b013e3181bfbf00. No abstract available. PMID 19901788
- [Background] Bendtsen TF, Moriggl B, Chan V, Borglum J. The Optimal Analgesic Block for Total Knee Arthroplasty. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):711-719. doi: 10.1097/AAP.0000000000000485. PMID 27685346
- [Background] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608
- [Background] Pert CB, Snyder SH. Properties of opiate-receptor binding in rat brain. Proc Natl Acad Sci U S A. 1973 Aug;70(8):2243-7. doi: 10.1073/pnas.70.8.2243. PMID 4525427
- [Background] Wang JK, Nauss LA, Thomas JE. Pain relief by intrathecally applied morphine in man. Anesthesiology. 1979 Feb;50(2):149-51. doi: 10.1097/00000542-197902000-00013. No abstract available. PMID 373503
- [Background] Meylan N, Elia N, Lysakowski C, Tramer MR. Benefit and risk of intrathecal morphine without local anaesthetic in patients undergoing major surgery: meta-analysis of randomized trials. Br J Anaesth. 2009 Feb;102(2):156-67. doi: 10.1093/bja/aen368. PMID 19151046
- [Background] Slappendel R, Weber EW, Dirksen R, Gielen MJ, van Limbeek J. Optimization of the dose of intrathecal morphine in total hip surgery: a dose-finding study. Anesth Analg. 1999 Apr;88(4):822-6. doi: 10.1097/00000539-199904000-00026. PMID 10195531
- [Background] Murphy PM, Stack D, Kinirons B, Laffey JG. Optimizing the dose of intrathecal morphine in older patients undergoing hip arthroplasty. Anesth Analg. 2003 Dec;97(6):1709-1715. doi: 10.1213/01.ANE.0000089965.75585.0D. PMID 14633547
- [Background] Choi S, Trang A, McCartney CJ. Reporting functional outcome after knee arthroplasty and regional anesthesia: a methodological primer. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):340-9. doi: 10.1097/AAP.0b013e318295d973. PMID 23788070
- [Result] The impact of arthritis in Canada: Today and Over the next 30 years. Arthritis Alliance of Canada. 2011 report.
- [Result] Hip and Knee Replacements in Canada. 2006 Report. Canadian Institute for Health Information(CIHI), Canadian Joint Replacement Registry